CLINICAL TRIAL: NCT04091425
Title: A Phase 1b Randomized, Double-blind, Placebo-Controlled, Crossover Study of 2 Single Intravenous Infusion Doses of TAK-925 in Subjects With Obstructive Sleep Apnea Who Are Experiencing Excessive Daytime Sleepiness Despite Adequate Use of CPAP
Brief Title: Study of TAK-925 in Participants With Obstructive Sleep Apnea (OSA) Who Are Experiencing Excessive Daytime Sleepiness (EDS) Despite Adequate Use of Continuous Positive Airway Pressure (CPAP)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Millennium Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TAK-925-2001
Record Dates: First submitted 2019-09-13; First posted 2019-09-16 (Actual); Last update posted 2020-04-20 (Actual); Status verified 2020-04

CONDITIONS: Obstructive Sleep Apnea
Keywords: Drug therapy
MeSH Terms: conditions — Sleep Apnea, Obstructive | interventions — TAK-925

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- TAK-925 Dose A (Experimental): TAK-925 dose A intravenous (IV) infusion in each treatment sequence (crossover design).
  Interventions: Drug: TAK-925
- TAK-925 Dose B (Experimental): TAK-925 dose B IV infusion in each treatment sequence (cross over design).
  Interventions: Drug: TAK-925
- Placebo (Placebo Comparator): TAK-925 placebo-matching IV infusion in each treatment sequence (crossover design).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: TAK-925 — TAK-925 IV infusion
  Arms: TAK-925 Dose A; TAK-925 Dose B
Drug: Placebo — TAK-925 placebo-matching IV infusion
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of administering a single intravenous (IV) infusion dose of TAK-925 to adults with obstructive sleep apnea (OSA) who are experiencing excessive daytime sleepiness (EDS) despite adequate use of CPAP as the primary OSA therapy.

DETAILED DESCRIPTION:
The drug being tested in this study is called TAK-925. TAK-925 is being tested to treat participants who have EDS due to OSA despite using CPAP. The study will evaluate the pharmacokinetics (PK), pharmacodynamics (PD), safety, and tolerability of a single IV dose of TAK-925 in participants with OSA.

The study will enroll approximately 42 patients. The study will utilize a three-way cross over design with a 24 hour wash-out between each treatment.

On Day 1 of each treatment period, TAK-925 or placebo will be administered as a single 9-hour IV infusion.

The multi-center study will be conducted in United States. The patient's participation in the study will last for up to 43 days and include an 8-day stay in the study clinic and a safety follow-up phone call 7 days after the end of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Has OSA diagnosed according to the international classification of sleep disorders-3 (ICSD-3) criteria and with current use of CPAP.
* Has a complaint of EDS despite "consistent use" of CPAP as defined by machine tracking time as having at least 4 hours of CPAP use/night on at least 70% during the approximately 1 month before randomization.
* If taking a stimulant medication for the treatment of excessive daytime sleepiness must be willing to discontinue medication before randomization into the study.
* Has a regular bedtime between 21:00 and 24:00 as verified by history and regular time in bed averaging between 7.5 and 9.0 hours/night and gets at least 6.5 hours/night on average of sleep, as defined by approximately 7 days of actigraphy supported by a sleep diary, which are completed at least 1 week before Study Day-2.
* Has a Epworth sleepiness scale (ESS) score of ≥10 at screening and Study Day -2, with or without stimulants.
* Nocturnal polysomnography (NPSG) demonstrates that the participant does not have other comorbid sleep disorders or clinically significant nocturnal hypoxemia (O2 saturation ≤80% for ≥5% of total sleep time) and that their apnea-hypopnea index (AHI) is ≤10.
* Has an average (of 4 sessions) baseline MWT sleep latency less than or equal to 20 minutes and no single session has a sleep latency of greater than 30 minutes as determined by the site investigator.

Exclusion Criteria:

* Has supine or standing average systolic blood pressure (SBP) ≥140 millimeters of mercury (mm Hg) or average diastolic blood pressure (DBP) ≥90 mm Hg at screening or Study Day-2; blood pressures will be averaged over 3 readings done 10 minutes (min) apart.
* A screening electrocardiogram (ECG) reveals a QT interval with Fridericia correction method >450 milliseconds (ms) (men) or >470 ms (women).
* Has a usual bedtime later than 01:00 or an occupation requiring nighttime shift work or variable shift work within the past 6 months or travel with significant jet lag within 14 days before Study Day-2.
* Short sleepers with chronic sleep deprivation who get on average less than 7.5 hours/night time in bed and/or less than 6.5 hours of sleep per night as defined by approximately 1 week of nocturnal actigraphy testing and supported by a sleep diary, both of which are completed at least 1 week before Study Day -2 admission to the clinical unit.
* Has a history of a sleep disorder other than OSA that is associated with EDS on the basis of interviews at the screening visit, such as, for example, restless legs syndrome, confirmed by prior pretreatment polysomnography (PSG) data demonstrating periodic limb movement during sleep (PLMS) >15.
* Has used any over-the-counter (OTC) or prescription medications with stimulating properties within 7 days before dosing or 5 half-lives (whichever is longer) that could affect the evaluation of EDS or any use of sodium oxybate within 3 months of screening.
* Has nicotine dependence that is likely to have an effect on sleep (e.g., a participant who routinely awakens at night to smoke) or challenge the conduct of this study (smokes ≥10 cigarettes/day) and/or the participant is unwilling to discontinue all smoking and nicotine use during the study.
* Has a caffeine consumption of more than 600 mg/day for 7 days before Study Day-1 (1 serving of coffee is approximately equivalent to 120 mg of caffeine).
* History or presence of any acutely unstable medical condition, behavioral or psychiatric disorder (including active suicidal ideation), or surgical history that could affect the safety of the subject or interfere with study efficacy, safety, PK assessments, or the ability of the subject to complete the study per the judgment of the investigator.

Ages: 18 Years to 67 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2019-11-21 (Actual); Primary Completion 2020-04-02 (Actual); Study Completion 2020-04-02 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants who Experience at Least One Treatment Emergent Adverse Event (TEAE) | Up to approximately 43 days
  An Adverse Event (AE) is defined as any untoward medical occurrence in a clinical investigation participant administered a drug; it does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (example, a clinically significant abnormal laboratory finding), symptom, or disease temporally associated with the use of a drug, whether or not it is considered related to the drug. A TEAE is defined as an AE with an onset that occurs after receiving study drug.
Percentage of Participants who Meet the Markedly Abnormal Criteria for Clinical Safety Laboratory Tests at Least Once Post a Regimen | Up to approximately 43 days
  Clinical laboratory evaluations include hematology, blood chemistry, and urinalysis.
Percentage of Participants who Meet the Markedly Abnormal Criteria for Vital Sign Measurements at Least Once Post a Regimen | Up to approximately 43 days
  Vital signs include heart rate, respiratory rate, systolic blood pressure (SBP) and diastolic blood pressure (DBP).
Percentage of Participants who Meet the Markedly Abnormal Criteria for 12-Lead Safety Electrocardiogram (ECG) Parameters at Least Once Post a Regimen | Up to approximately 43 days
  A standard 12-lead ECG will be performed.

SECONDARY OUTCOMES:
Ceoi: Observed Plasma Concentration at the end of Infusion for TAK-925 | Pre-dose, at multiple time points (up to 9 hours) after start of infusion, and at multiple time points (up to 15 hours) after end of infusion on Day 1 each Treatment Period
AUC∞: Area Under the Plasma Concentration-Time Curve From Time 0 to Infinity for TAK-925 | Pre-dose, at multiple time points (up to 9 hours) after start of infusion, and at multiple time points (up to 15 hours) after end of infusion on Day 1 each Treatment Period
AUClast: Area Under the Plasma Concentration-Time Curve from Time 0 to Time of the Last Quantifiable Concentration for TAK-925 | Pre-dose, at multiple time points (up to 9 hours) after start of infusion, and at multiple time points (up to 15 hours) after end of infusion on Day 1 of each Treatment Period

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Takeda
Locations (18):
- United States (18):
  - Wright Clinical Research, Alabaster, Alabama
  - Pulmonary Associates Clinical Trials, Glendale, Arizona
  - Preferred Research Partners, Inc., Little Rock, Arkansas
  - Stanford School of Medicine, Redwood City, California
  - Pacific Research Network, Inc, San Diego, California
  - Delta Waves Sleep Disorders and Research Center, Colorado Springs, Colorado
  - MD Clinical, Hallandale, Florida
  - Research Centers of America, Hollywood, Florida
  - Jacksonville Center for Clinical Research, Jacksonville, Florida
  - Pulmonary Disease Specialists, PA, d/b/a PDS Research, Kissimmee, Florida
  - Florida Pulmonary Research Institute, LLC, Winter Park, Florida
  - NeuroTrials Research, Inc., Atlanta, Georgia
  - SleepCare Research Institute, Inc. d/b/a Clinical Research Institute, Stockbridge, Georgia
  - Helene A. Emsellem, MD PC trading as "The Center for Sleep & Wake Disorders", Chevy Chase, Maryland
  - CTI Clinical Trial and Consulting Services, Cincinnati, Ohio
  - The Cleveland Clinic Foundation, Cleveland, Ohio
  - Bogan Sleep Consultants, LLC, Columbia, South Carolina
  - Sleep Therapy & Research Center, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: Yes
Takeda makes patient-level, de-identified data sets and associated documents available for all interventional studies after applicable marketing approvals and commercial availability have been received (or program is completely terminated), an opportunity for the primary publication of the research and final report development has been allowed, and other criteria have been met as set forth in Takeda's Data Sharing Policy (see www.TakedaClinicalTrials.com for details). To obtain access, researchers must submit a legitimate academic research proposal for adjudication by an independent review panel, who will review the scientific merit of the research and the requestor's qualifications and conflict of interest that can result in potential bias. Once approved, qualified researchers who sign a data sharing agreement are provided access to these data in a secure research environment.